CLINICAL TRIAL: NCT02131948
Title: Regulation of Endogenous Glucose Production by Brain Insulin Action
Acronym: Nasal insulin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REB 12-5032A
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Insulin Resistance, Diabetes
Keywords: Insulin resistance; Brain insulin action; Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal insulin (Experimental): 40 IU of intranasal insulin
  Interventions: Drug: Intranasal insulin
- Intranasal placebo (Placebo Comparator): Placebo comparator to intranasal insulin
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal insulin — Intranasal spray
  Other Names: Humalog lispro 40 IU intranasally
  Arms: Intranasal insulin
Drug: Intranasal placebo — Intranasal spray
  Other Names: Diluent intranasally
  Arms: Intranasal placebo

SUMMARY:
It is well known that the hormone insulin lowers blood glucose in part by acting directly on the liver and reducing hepatic glucose production. Animal studies have shown that the hormone insulin can act on the brain to indirectly lower glucose production by the liver. We aim to test whether this is true in humans by giving insulin intranasally. It has previously been shown that a nasal spray can deliver insulin directly to the brain without affecting circulating insulin concentration.

DETAILED DESCRIPTION:
Each study participant will be admitted to hospital the evening prior to the study. Following admission each study participant will be provided with a standardized dinner. At 7am (t=0) the next day we will begin a primed, constant intravenous infusion d2 glucose (a stable isotope of glucose, the enrichment of which can be measured by gas chromatography mass spectrometry, allowing us to calculate endogenous glucose production rates) and continue this for 8 hours. At the same time (7am) a pancreatic clamp will be started as described above for 8 hours. Blood samples will be analysed with a glucometer for instant blood glucose readings At 9 am (+120 minutes) intranasal placebo or insulin will be administered. The insulin (Humalog Lispro 100 IU/ml, Eli Lily, Canada) and placebo (diluent) will be transferred to a metered nasal device (Pharmasystems, Ontario UPC: 063636 802721, Item 10271) immediately prior to use. This device dispenses 0.1ml (10 IU) per puff. 4X0.1 ml puffs/vials (2 per nostril) will be administered at rate of 2 (one in each nostril) every 60 seconds. Blood will be drawn at t=0, 30, 60, 120 and every 10 minutes thereafter for 6 hours. In order to match peripheral lispro concentrations between study visits, a small dose of Humalog (lispro) insulin will be administered intravenously at 9am, during the placebo arm of the study. Based on the pharmacokinetics of Humalog lispro (personal communication from Eli Lilly), we propose to administer 0.005 IU/kg over 30 minutes. 20% dextrose will be administered to maintain euglycemia as necessary. Insulin, glucagon, and glucose isotopic enrichment will be measured. The enrichment data and glucose infusion will be used to calculate steady state glucose production.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 60 years
2. Body mass index 20-27.
3. Hemoglobin in the normal range.
4. Normal glucose tolerance in response to a 75g, 2-hr oral glucose tolerance test
5. Women of reproductive age should be on contraception (oral contraceptive pill or intra-uterine device/coil) for at least 2 months prior to and after the study.

Volunteers who have taken part in the study with the previously approved protocol will be eligible to participate in the amended study, if they provide their informed consent

Exclusion Criteria:

Study participant with a history of hepatitis/hepatic disease that has been active within the previous two years.

2. Any current or previous history of biliary disease (including gall stones, biliary atresia and cholecystitis) or pancreatitis.

3. Any current or previous history of endocrine disease, dyslipidemia or malignancy 4. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL) genitourinary, hematological systems, or has severe uncontrolled treated or untreated hyper/ hypotension (sitting diastolic BP > 100 or systolic > 180 or systolic BP<100) or proliferative retinopathy 5. Use of immunosuppressive agents at any time during the study 6. Allergy to any study medication 7. Pregnancy or breastfeeding 8. Heavy smoker 9. Prior nasoduodenal tube insertion under fluoroscopic guidance. 10. Fasting blood glucose > 6.0 mmol/l or known diabetes. 11. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.

12. Any nasal pathology likely to affect absorption of insulin or insertion of nasoduodenal tube.

13. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH > 6 mU/l 14. Current addiction to alcohol or substances of abuse as determined by the investigator.

15. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation 16. Taking any regular prescription or non-prescription medications at the time of the study. Occasional use of medications such as acetoaminophen or Tylenol 1 or any use of natural health products may be permitted at the discretion of the investigator.

17. Will not donate blood three months prior to and three months post study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Endogenous glucose production | 8 hours
  Effects of intranasal insulin and placebo on endogenous glucose production will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Tornto General Hospital, UHN, Toronto, Ontario, Canada